CLINICAL TRIAL: NCT05604300
Title: Effectiveness of Vitamin E Incorporated Oat Supplementation in Metabolic Syndrome
Brief Title: The Role of Vitamin E Incorporated Oat Supplementation in Metabolic Syndrome (MetS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Gold Choice Food Industries Sdn. Bhd (Unknown)
Responsible Party: Principal Investigator, Dr. Lee Lai Kuan, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: USM/JEPeM/22020101
Record Dates: First submitted 2022-10-27; First posted 2022-11-03 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin E incorporated oat (Active Comparator): Oral vitamin E incorporated oat supplementation
  Interventions: Dietary Supplement: Vitamin E incorporated oat supplement
- Placebo (Placebo Comparator): Oral oat supplementation
  Interventions: Dietary Supplement: Oat supplement
- Control (No Intervention): Control

INTERVENTIONS:
Dietary Supplement: Vitamin E incorporated oat supplement — A twice daily supplementation of Vitamin E incorporated oat for 12 weeks
  Arms: Vitamin E incorporated oat
Dietary Supplement: Oat supplement — A twice daily supplementation of oat for 12 weeks
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effect of vitamin E incorporated oat supplementation among the metabolic syndrome (MetS) patients.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is a common metabolic disorder, characterized by a cluster of cardiovascular disease (CVD) risk factors including elevated blood glucose level, dyslipidemia, abdominal obesity, and high blood pressure. It was initially introduced by WHO in 1998 as insulin resistance, in addition to two other risk factors, being prerequisites for diagnosis. Other criteria, such as the National Cholesterol Education Program Expert Panel III (ATP III) and the International Diabetes Federation, were later established to improve the diagnosis of MetS. In the new global economy, MetS has become a central issue for public health concern due to the parallel increase in diabetes, CVD, and obesity. Clinical and epidemiological data have indicated that metabolic syndrome starts with central obesity. Since the global incidence of obesity has doubled in the last 30 years, the prevalence of metabolic syndrome has also increased exponentially. Therefore, obesity has been seen to be the primary cause of the metabolic syndrome since it significantly relates to all metabolic risk factors. It was estimated that in 2017, there were 451 million people with diabetes worldwide and is expected to reach 693 million by 2045. Primarily, almost half of the people (49.7%) is estimated to be living with undiagnosed diabetes. These figures signify that obesity and insulin resistance is recognized as the primary pathophysiology underlying metabolic syndrome. Lifestyle intervention including diet control is recommended as the fundamental approach for all patients with metabolic syndrome. One of the discussed components was the potential role of oat-containing beta-glucan in the prevention of metabolic syndrome. The general principle of dietary provision for CVD is by providing a 3-5 serving of whole grain per day throughout the intervention trial. The European

Food Safety Authority gave a favorable view on the health claim for foods containing oat beta glucan:

"Regular consumption of oat b-glucans can actively lower/reduce blood LDL cholesterol and total cholesterol". Despite a large body of studies demonstrating the association between oat consumption and cardiovascular disease, limited information from clinical trials is available on the effective doses of whole-grain consumption on metabolic control. However, it is debatable if a higher provision of whole-grain consumption confers beneficial effects on metabolic syndrome and cardiovascular disease. β-glucan is the most abundant soluble fibre in oats and barley. It has been shown to lower serum cholesterol and improve postprandial insulin and glucose responses in healthy and 3 diabetic adult. While dietary fibre is by far the most essential nutritional feature of whole grains, they also contain a variety of phytochemicals that may have therapeutic metabolic benefits. Alkylresorcinols, flavonoids, lignans, phenolic acids, phytosterols, and tocols (tocopherols and tocotrienols) are among some of the phytochemicals located principally in the outer bran layer. It has been proposed that these and other health benefits of whole grains may be due to a synergistic action of fibre and phytochemical constituents. Furthermore, more studies have suggested a dietary intervention of bioactive enriched as functional foods for adults at risk of metabolic syndrome. However, limited studies have been exploring high fiber consumption and antioxidant properties as distinct and separate dietary management; thus the effectiveness of collective management is not being explored adequately. Furthermore, prospective studies that have examined this association are scarce. Bioactive components have been proposed to confer benefits to reduce the consequential of oxidative stress. Antioxidants, especially the tocotrienols, are among novel compounds studied extensively for their metabolic effects. Tocotrienol, a functional nutritional component exhibiting anti-inflammatory, antioxidant, and cell signaling-mediating properties, could be helpful as an adjuvant treatment for obesity and diabetes diseases. Tocotrienol has been shown to have potent anti-inflammatory and anti-cancer properties by modifying multiple molecular signaling pathways that are usually unaffected by tocopherol. Tocotrienol, particularly γ-tocotrienol lowers the incidence of cardiovascular disease, diabetes, and metabolic syndrome. Moreover, emerging data indicate that tocotrienol is a promising anti-obesity agents by reducing body weight and improve plasma glucose and lipid hepato-protective effects in individuals with nonalcoholic fatty liver disease which is a complication associated with obesity.

Previous study has demonstrated a lower bioavailability of vitamin E among metabolic syndrome patients. This perturbing condition spiked the interest of researchers in incorporating vitamin E in diet modulation. In addition, the lack of studies in MetS people taking vitamin E in typical dietary amounts makes it difficult to make specific nutritional tocotrienol recommendations for this group. Thus, study of tocotrienol pharmacokinetics in MetS is needed and the identification of low-energy, nutrient-dense dietary methods to improve vitamin E status. to search for some potential complementary medicine to combat MetS. The use of oat as food source as part of the dietary regimen, or functional food to alleviate the disease progression is the novel research focus among the scientific communities. However, limited studies have been strategized to outline the efficacy of incorporating vitamin E into functional foods for the amelioration of chronic disease. With the aforementioned, this randomised, placebo-controlled, double-blinded human clinical trial is aimed to determine the efficacy of 12 weeks supplementation of vitamin E incorporated oat products as part of the dietary regimen among the MetS individuals. Secondary and tertiary outcomes include the assessment of circulating antioxidative status and oxidative stress level, inflammatory markers, nutritional status and quality of life. The compliancy and tolerability of the supplementation will be assessed periodically.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old and above
2. Individuals who have been identified as having metabolic syndrome (meet ≥3 out of 5 NCEP-ATP III Criteria)
3. Stable weight (± 2 kg during the past 3months) to ensure reliable weight changes with the treatment given.
4. Not taking antioxidant/anti-inflammatory supplements (Example of antioxidant: vitamin C, vitamin E, grape seed extract, garlic capsule, ginkgo biloba); (Example of the anti-inflammatory supplement: fish oil, curcumin extract, ginger extract, spirulina)

Exclusion Criteria:

1. Having liver (chronic liver failure, cirrhosis, all types of hepatitis), kidney (chronic kidney disease, haemodialysis) or haematological (anaemia, thalassemia, haemophilia) disorders
2. Cancer (all types) and endocrine disorders (Cushing's disease, gigantism and hyperthyroidism).
3. Alcohol and drug abuse (self-mentioned or as recorded in the medical card)
4. Hormone replacement therapy (for at least three months prior to entering the study)
5. Use of steroids, chemotherapy, immunosuppressant, or radiotherapy
6. Currently pregnant or lactating
7. Participations currently under another supplementary program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Triacylglycerol concentrations | Baseline and 12 weeks
  Triacylglycerol concentration is measured in mg/dL
Change in HDL-cholesterol concentrations | Baseline and 12 weeks
  HDL-cholesterol concentration is measured in mg/dL
Change in fasting blood glucose concentrations | Baseline and 12 weeks
  Fasting blood glucose concentration is measured in mg/dL
Change in systolic and diastolic blood pressure | Baseline and 12 weeks
  Systolic and diastolic blood pressure are measured in mmHg
Change in waist circumference | Baseline and 12 weeks
  Waist circumference is measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: Lai Kuan Lee, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Advanced Medical and Dental Institute (AMDI), Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No